CLINICAL TRIAL: NCT07126951
Title: A Pragmatic Randomized Controlled Pilot Clinical Trial of Ultrasound Guiding Pharmacopuncture Therapy for Acute Low Back Pain Following Traffic Accidents
Brief Title: Pilot Study: Clinical Trial of Ultrasound Guiding Pharmacopuncture Therapy for Acute Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2025-08
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain (LBP)
Keywords: pharmacopuncture; Ultrasound Guiding
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: A Pragmatic randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided Deep Pharmacopuncture Treatment (Experimental): Participants in this arm will receive integrative Korean medicine treatment combined with ultrasound-guided deep pharmacopuncture. The integrative treatment includes acupuncture, Chuna manual therapy (focused on cervical and lumbar regions), and oral herbal medicine administered during hospitalization.
  In addition to these treatments, patients in this group will receive ultrasound-guided pharmacopuncture therapy once daily from Day 2 to Day 4 of hospitalization, for a maximum of three sessions. The pharmacopuncture procedure involves injecting 4 cc of herbal extract into deep lumbar tissue using a 26G sterile needle under real-time ultrasound guidance. The target site is selected based on lumbar spine X-ray findings (disc narrowing) and patient-reported radiating pain. The needle is inserted using an in-plane approach to visualize the needle tip reaching the posterior facet joint of the most symptomatic lumbar segment.
  Interventions: Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group were received Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Ultrasound-guided Deep Pharmacopuncture Treatment; Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Ultrasound-guided Deep Pharmacopuncture Treatment — Participants in this group will receive ultrasound-guided deep pharmacopuncture in addition to integrative Korean medicine treatment (acupuncture, herbal medicine, and Chuna therapy). The pharmacopuncture involves injecting 4 cc of herbal extract into deep lumbar tissues, targeting the posterior facet joint of the most symptomatic segment.
  Using a real-time ultrasound-guided in-plane technique, the needle path and tip are visualized to ensure accurate and safe delivery. Treatment is administered once daily for up to 3 days (hospital Days 2-4).
  This intervention differs from conventional methods by using ultrasound to guide precise, deep-tissue injection, enhancing both safety and treatment accuracy.
  Arms: Korean medical treatment
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This pilot randomized controlled clinical trial aims to evaluate the effectiveness and safety of ultrasound-guided deep pharmacopuncture therapy for acute low back pain (LBP) that occurs within seven days following a traffic accident. While traditional Korean medicine-including acupuncture, herbal medicine, pharmacopuncture, and Chuna manual therapy-is commonly used for post-accident injuries, few studies have focused on deep pharmacopuncture administered under ultrasound guidance. This study will provide preliminary evidence to assess whether ultrasound-guided techniques offer added clinical benefits.

A total of 40 patients hospitalized at Jaseng Hospital of Korean Medicine in Haeundae, Korea, will be recruited and randomly assigned into two groups: the intervention group will receive integrative Korean medicine therapy plus ultrasound-guided pharmacopuncture, while the control group will receive integrative Korean medicine therapy alone. Both groups will undergo treatment during hospitalization, with the pharmacopuncture administered up to three times between hospital day 2 and day 4 in the intervention group. Baseline assessment will be done on day 2 before treatment, and the primary outcome will be measured on day 5. Follow-up assessments will be conducted at 2 and 4 weeks via telephone.

The primary outcome is the change in low back pain intensity as measured by the Numeric Rating Scale (NRS). Secondary outcomes include radiating pain, lumbar range of motion, Oswestry Disability Index (ODI), EQ-5D for quality of life, and the Patient Global Impression of Change (PGIC). Adverse events will also be monitored and classified according to established safety criteria.

This study will utilize both intention-to-treat (ITT) and per-protocol (PP) analyses, with linear mixed models and multiple imputation used to address missing data. Given the limited existing evidence on ultrasound-guided deep pharmacopuncture, this trial is designed to explore its feasibility and provide the groundwork for future large-scale trials.

Participants will be selected based on strict inclusion and exclusion criteria to ensure safety and consistency. Ethical standards including informed consent, data privacy, and ongoing safety monitoring will be rigorously upheld throughout the study.

DETAILED DESCRIPTION:
This pragmatic, randomized, controlled pilot study investigates the comparative clinical effectiveness and safety of ultrasound-guided deep pharmacopuncture versus conventional integrative Korean medicine treatment for acute low back pain (LBP) occurring within 7 days after a traffic accident.

The study will enroll 40 hospitalized patients aged 19-70 who report moderate to severe acute LBP (NRS ≥5) and have disc narrowing visible on lumbar X-rays. Participants will be randomly assigned to one of two treatment arms (n=20 per group) using a block randomization procedure. The trial will proceed through a screening/enrollment phase, active inpatient treatment, and follow-up evaluations at 2 and 4 weeks post-enrollment.

The intervention group will receive a combination of standard integrative Korean medicine treatment and 1 to 3 sessions of ultrasound-guided deep pharmacopuncture between hospital day 2 and 4. The control group will receive standard care only, which includes acupuncture, non-ultrasound-guided pharmacopuncture, herbal medicine, and Chuna manual therapy.

The primary outcome is change in low back pain intensity (NRS) from baseline (Day 2 pre-treatment) to Day 5. Secondary outcomes include radiating pain, lumbar range of motion (ROM), functional status (Oswestry Disability Index), quality of life (EQ-5D-5L), and overall improvement (Patient Global Impression of Change). Adverse events will be systematically monitored and assessed.

The trial is designed to evaluate the feasibility, effect size estimation, and safety profile of ultrasound-guided pharmacopuncture in preparation for a larger-scale confirmatory trial. Analyses will follow both ITT and PP principles, with linear mixed models and imputation techniques for handling missing data.

The study adheres to ethical guidelines, including informed consent, privacy protection, and safety monitoring. Monitoring will be conducted by third parties per KCGP standards to ensure data quality and patient protection.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

Adults aged 19 to 70 years.

Patients who developed acute low back pain within 7 days after a traffic accident.

Numeric Rating Scale (NRS) score of 5 or higher for low back pain.

Radiological evidence of disc narrowing on lumbar spine X-ray.

Complaints of radiating leg pain.

Hospitalized for treatment related to the traffic accident.

Able and willing to provide written informed consent voluntarily.

Exclusion Criteria:

Participants will be excluded if they meet any of the following:

Diagnosed with serious underlying conditions causing back pain (e.g., malignancy, spinal infection, inflammatory spondylitis).

Presence of progressive or severe neurological deficits.

Underwent lumbar surgery or procedures within the past 3 weeks.

Back pain caused by non-spinal soft tissue disorders (e.g., fibromyalgia, rheumatoid arthritis, gout).

Presence of chronic conditions that could interfere with study results (e.g., cardiovascular disease, renal disease, diabetic neuropathy, dementia, epilepsy).

Taking medications that could affect study outcomes (e.g., steroids, immunosuppressants, psychiatric drugs).

Contraindicated or unsafe for acupuncture (e.g., bleeding disorders, anticoagulant therapy, severe diabetes with infection risk, severe cardiovascular conditions).

Currently pregnant or planning pregnancy.

Diagnosed with severe mental illness.

Participation in other clinical trials (excluding observational studies).

Unable to properly complete the informed consent form.

Deemed inappropriate for participation by the investigator for any other reason.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Low back Pain intensity scale: Numeric Rating Scale(NRS) | Day1, Baseline(day2), day3, day4, day5, 2week after enrollment, 4week after enrollment
  The NRS is a numeric scale used to quantify the patient's subjective experience of pain. Patients rate their current low back pain on a scale from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable.

SECONDARY OUTCOMES:
Radiating pain intensity scale: Numeric Rating Scale(NRS) | Day1, Baseline(day2), day3, day4, day5, 2week after enrollment, 4week after enrollment
  This scale assesses the severity of radiating pain (e.g., pain extending to the legs). Patients rate their current radiating pain on a 0-10 scale, where 0 indicates no pain and 10 indicates the worst possible radiating pain.
Oswestry Disability Index (ODI) | Baseline(day2), day5, 2week after enrollment, 4week after enrollment
  The ODI is used to assess functional impairment due to low back pain. It consists of 10 items, each scored from 0 to 5, for a maximum score of 50. The final score is calculated as the average of the answered items and reflects the patient's level of disability in daily life.
EuroQol-5D-5L (EQ-5D) | Baseline(day2), day5, 2week after enrollment, 4week after enrollment
  EQ-5D is a standardized tool for measuring health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on five levels (1 = no problem, 5 = extreme problem). A Korean-specific value set will be applied to calculate utility scores.
Physical Examination - Lumbar Active Range of Motion (AROM) | Baseline(day2), day3, day4, day5
  This measures the maximum range of motion in the lumbar spine that the patient can achieve without pain. Six movements are assessed: flexion, extension, left and right lateral bending, and left and right rotation. Measurements are taken using a goniometer. If the patient refuses due to severe pain, the result is recorded as 0 degrees.
Patient Global Impression of Change (PGIC) | day5, 2week after enrollment, 4week after enrollment
  PGIC is a 7-point scale where patients rate their overall improvement following treatment, ranging from "very much improved" to "very much worse."
Adverse Events (AE) | Baseline(day2), day3, day4, day5, 2week after enrollment, 4week after enrollment
  Any unfavorable and unintended sign, symptom, or disease temporally associated with the treatment will be recorded, regardless of a causal relationship. Events will be monitored and classified by severity (mild, moderate, severe) using Spilker's criteria, and by causality using a 6-point WHO-UMC scale.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Haeundae, Jaseng Hospital of Korean Medicine, South Korea

IPD SHARING:
Plan to Share IPD: No